CLINICAL TRIAL: NCT03837158
Title: Is the Stabilization of a Mandibular Overdenture Employing Four Novel One-piece Immediately Loaded TiZr Implants With Miniaturized Stud-type Attachments a Feasible Alternative to Two Two-piece Early Loaded Tissue-level Implants With Regular Stud-type Attachments?
Brief Title: Titanium Zirconium (TiZr) Mini Implants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mini 1286_2018
Record Dates: First submitted 2019-01-30; First posted 2019-02-12 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Dental Implants
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-group (Experimental): Two Tissue Level TiZr Sand blasted long grit acid-etched (SLA) implants placed in positions 33 and 43 (diameter 3.3mm, length ≥10mm), early loading
  Interventions: Procedure: early loading
- Experimental-group (Experimental): Four narrow-diameter implants (NDI) TiZr SLA implants in positions 34, 32, 42, and 44 (diameter 2.4mm, length ≥10mm), immediate loading
  Interventions: Procedure: immediate loading

INTERVENTIONS:
Procedure: early loading — two TiZr implants on SLA surface
  Arms: Control-group
Procedure: immediate loading — four TiZr implants on SLA surface
  Arms: Experimental-group

SUMMARY:
H0: "Within the first year post-placement, four interforaminally placed, immediately loaded 2.4 mm narrow-diameter one-piece TiZr implants with miniaturized stud-type attachments show improved patient-reported outcome measures (PROMS) compared to two interforaminally placed, early loaded, TiZr two-piece implants with stud-type attachments to retain a mandibular overdenture."The specific aim is to compare both treatment alternatives to evaluate which one may be recommended for elderly edentulous patients.

ELIGIBILITY:
Inclusion Criteria:

* At patient level:

  * Written informed consent
  * Age ≥ 18 years
  * Sufficient complete dentures (Marxkors and Ferger, 1989) not older than 1 year
  * Patient is unsatisfied with mandibular denture to the degree that he/she seeks treatment
* At site level:

  * Healed edentulous mandible (minimum 8 weeks since last extraction)
  * Minimal ridge dimensions 5.5 mm (width) by 12 mm (height) in the anterior (interforaminal) area, allowing the placement of 3.3 (endosseous diameter) by 10 mm (length) implants
  * Opposing dentition: complete denture on a edentulous maxilla
  * Physical status (PS) 1 and 2 (American Society of Anesthesiologists)

Exclusion Criteria:

* At patient level

  * Any physical or mental disorder that would interfere with the ability to perform adequate oral hygiene or the capability of providing written informed consent and compliance to the protocol
  * Any disorder that would interfere with wound healing or represent a contraindication for oral surgery such as, but not limited to, uncontrolled diabetes or conditions resulting in or requiring immunosuppression, radiation, chemotherapy, frequent use of antibiotics or antiresorptive medication such as bisphosphonates
  * Pregnancy or lactation
  * Heavy smoking habit with > 20 cig/d
  * Severe bruxism or clenching habits, present oro-facial pain
* At site level:

  * Ridge defects requiring staged bone augmentation procedures (simultaneous Guided Bone Regeneration (GBR) within the ridge contour allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2033-08 (Estimated)

PRIMARY OUTCOMES:
Geriatric Oral Health Assessment Index (GOHAI) | One-year follow-up
  Change from baseline questionnaires in Oral Health Related Quality of Life (OHRQoL).
  Scores 0-60: higher values represent lower OHRQoL

SECONDARY OUTCOMES:
Additional Oral Health Impact Profile for edentulism (OHIP-EDENT) | Follow-up (up to 365 days)
  Change from baseline questionnaires
Additional PROM Denture Satisfaction Index (DSI) | Baseline, follow-up (up to 365 days)
  Change in Denture Satisfaction higher values represent better satisfaction (0-1200mm)
Implant Survival | at implant loading (at 24 hours for arm B, at 6-8 weeks for arm A), at the one-year follow-up
  Survival (yes/no)
Implant Success | at implant loading (at 24 hours for arm B, at 6-8 weeks for arm A), at the one-year follow-up
  Success according to Misch (2007) Misch criteria scores 1-4: higher values represent better success
Prosthetic Survival | Baseline, follow-up (up to 365 days)
  Prosthetic Survival (yes/no): is the denture still in place?
Chewing Efficiency | Baseline, follow-up (up to 365 days)
  Color mixing test
Plaque Index | at implant loading (at 24 hours for arm B, at 6-8 weeks for arm A), at the one-year follow-up
  Plaque Index Scores 0-3 3= thick plaque is visible along gingival margin 2= plaque is visible along gingival margin, with or without air drying
  1= following air drying, plaque is not visible but can be wiped off with an explorer 0= following air drying, plaque is not visible nor can be wiped off with an explorer
Bleeding Index | at implant loading (at 24 hours for arm B, at 6-8 weeks for arm A), at the one-year follow-up
  Bleeding Index Scores 0-3 0= Healthy gingival
  1. Gingival look inflamed, but don't bleed when probed
  2. Gingival look inflamed and bleed when probed
  3. Ulceration and spontaneous bleeding
Pocket Probing depth | at implant loading (at 24 hours for arm B, at 6-8 weeks for arm A), at the one-year follow-up
  depth measured in mm
Time-Cost-Analysis | After surgery, after implants loading, after follow-up (up to 365 days)
  Total treatment time will be collected and added. Total treatment cost will be evaluated and a ratio will be calculated. The groups will be compared on the base of this ration
Cost Effectiveness and Willingness to Pay | Total change and time at 1y follow-up
  Cost effectiveness wil be calculated as a ratio of treatment cost in relation to change of GOHAI sum score. This will allow to evaluate how much monetary item is needed to achieve a change in GOHAI
In-vivo evaluated loss of retentive force | after implant loading (expected to be after 6 weeks on average) and at follow-up (up to 365 days)
  Measurement with a hand-held digital force gauge

CONTACTS AND LOCATIONS:
Overall Officials: Beat Wallkamm, Dr, Principal Investigator — Private Practice; Martin Schimmel, Prof, Study Director — University of Bern
Locations (2):
- Switzerland (2):
  - Private Practice Dr. B. Wallkamm, Langenthal, Canton of Bern
  - University of Bern, Bern

IPD SHARING:
Plan to Share IPD: No
It is not planned to use the data of this study for future research.